CLINICAL TRIAL: NCT02292368
Title: Neurological Effects of Acupuncture to Prevent Radiation-induced Xerostomia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2013-0769; 1R01CA148707 (NIH); NCI-2015-00350 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2014-11-10; First posted 2014-11-17 (Estimated); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Cancer; Xerostomia; Radiation-induced Xerostomia; Acupuncture; Nasopharyngeal cancer; Radiation therapy; XRT; Electroencephalogram; EEG; Xerostomia questionnaire; XQ; MD Anderson Symptom Inventory - Head & Neck; MDASI-HN; Questionnaires; Surveys
MeSH Terms: conditions — Head and Neck Neoplasms; Xerostomia; Nasopharyngeal Neoplasms | interventions — Surveys and Questionnaires; Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture - One Type (Experimental): Participants recruited between weeks 3-5 of radiotherapy. Acupuncture treatments given within 3 to 7 days of each other during Weeks 3-5 of regularly scheduled radiotherapy visits. It should take about 20 minutes to complete the acupuncture session each time.
  At each acupuncture session, 3 questionnaires completed before each session that ask about dry mouth, any other symptoms, and treatment expectations. It should take about 5 minutes total to complete these questionnaires. Participants also complete another brief questionnaire about dry mouth after each session. It should take about 1 minute to complete this questionnaire.
  Participants also have an EEG at each acupuncture treatment. EEG recorded 5 minutes before acupuncture, during acupuncture, and for 5 minutes after acupuncture. Total visit time will last about 45-60 minutes.
  Interventions: Behavioral: Questionnaires; Procedure: Acupuncture; Procedure: Electroencephalogram (EEG)
- Acupuncture - Different Type (Experimental): Participants recruited between weeks 3-5 of radiotherapy. Acupuncture treatments given within 3 to 7 days of each other during Weeks 3-5 of regularly scheduled radiotherapy visits. It should take about 20 minutes to complete the acupuncture session each time.
  At each acupuncture session, 3 questionnaires completed before each session that ask about dry mouth, any other symptoms, and treatment expectations. It should take about 5 minutes total to complete these questionnaires. Participants also complete another brief questionnaire about dry mouth after each session. It should take about 1 minute to complete this questionnaire.
  Participants also have an EEG at each acupuncture treatment. EEG recorded 5 minutes before acupuncture, during acupuncture, and for 5 minutes after acupuncture. Total visit time will last about 45-60 minutes.
  Interventions: Behavioral: Questionnaires; Procedure: Acupuncture; Procedure: Electroencephalogram (EEG)

INTERVENTIONS:
Behavioral: Questionnaires — At each acupuncture session, 3 questionnaires completed before each session that ask about dry mouth, any other symptoms, and treatment expectations. It should take about 5 minutes total to complete these questionnaires. Participants also complete another brief questionnaire about dry mouth after each session. It should take about 1 minute to complete this questionnaire.
  Other Names: Surveys
Procedure: Acupuncture — Acupuncture treatments given within 3 to 7 days of each other during Weeks 3-5 of regularly scheduled radiotherapy visits. It should take about 20 minutes to complete the acupuncture session each time.
Procedure: Electroencephalogram (EEG) — Participants have an EEG at each acupuncture treatment. EEG recorded 5 minutes before acupuncture, during acupuncture, and for 5 minutes after acupuncture. Total visit time will last about 45-60 minutes.
  Other Names: EEG

SUMMARY:
The goal of this clinical research study is to learn which areas of the brain respond to acupuncture that is designed to prevent xerostomia (dry mouth) in patients with head and neck cancer. Researchers also want to learn if acupuncture can help prevent dry mouth and improve patient quality of life.

DETAILED DESCRIPTION:
Dry mouth is a common problem in cancer patients who have received radiation treatment to the head and neck. Acupuncture is a technique that may treat symptoms by inserting very thin, solid, sterile, stainless steel needles into the skin at specific points.

Study Groups:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the flip of a coin) into 1 of 2 groups. You will have an equal chance of being in either group.

Group 1 will receive one type of acupuncture for one session and another type of acupuncture for the second session.

Group 2 will receive one type of acupuncture for one session and another type of acupuncture for the second session.

You will not know if you are assigned to Group 1 or Group 2.

Study Visits:

Your acupuncture treatments will be within 3 to 7 days of each other during Weeks 3-5 of your regularly scheduled radiotherapy visits. It should take about 20 minutes to complete the acupuncture session each time.

At each acupuncture session, you will complete 3 questionnaires before each session that ask about dry mouth, any other symptoms you may be having, and your treatment expectations. It should take about 5 minutes total to complete these questionnaires. You will also complete another brief questionnaire about dry mouth after each session. It should take about 1 minute to complete this questionnaire.

You will also have an EEG at each acupuncture treatment. The EEG will be recorded 5 minutes before acupuncture, during acupuncture, and for 5 minutes after acupuncture. Total visit time will last about 45-60 minutes.

You will give a saliva sample before and after each acupuncture treatment to measure the amount of saliva produced.

Length of Study:

You will remain on study for about 1 week. Your participation in the study will be over after you complete the dry mouth questionnaire after your second acupuncture session.

This is an investigational study.

Up to 50 patients will take part in this multicenter study. Up to 30 will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age and be able to give informed consent.
2. Diagnosed with head and neck cancer, which will be primarily nasopharyngeal, and scheduled to undergo IMRT or proton with or without concurrent chemotherapy at MD Anderson or Fudan University.
3. Treatment plan that includes external beam radiation at a mean dose of at least 24 Gy or more to one of the parotid glands (the other gland can receive less than 24 Gy).
4. Anatomically intact parotid and submandibular glands.
5. Karnofsky performance status > 60.
6. Must be right-handed.

Exclusion Criteria:

1. History of xerostomia prior to head and neck radiation therapy or history of Sjögren's disease or another underlying systemic illness known to cause xerostomia.
2. Prior head and neck radiation treatment.
3. Suspected or confirmed physical closure of salivary gland ducts on either side.
4. Known bleeding disorders or taking any dose of warfarin or heparin.
5. Upper or lower extremity deformities (ie, missing limbs or scars that prevent needle insertion at the acupuncture points) that could interfere with accurate acupoint location or alter the energy pathway as defined by traditional acupuncture theory.
6. Local skin infections at or near the acupuncture sites or are under treatment for active systemic infection.
7. History of cerebrovascular accident or spinal cord injury since the mechanism of acupuncture may be associated with central nervous system activity.
8. Documented history of mental incapacitation or significant emotional or psychiatric disorder (i.e. bipolar, schizophrenia) that, in the opinion of the investigator, precludes study entry as these patients may not be able to cooperate with this slightly invasive procedure or with the data collection process.
9. Current acknowledged use of any illicit drugs or evidence of alcohol abuse as defined by The American Psychiatric Association criteria.
10. Patients who are currently receiving acupuncture for any condition or if they have ever had acupuncture before.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-11-10 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Relative Changes of EEG Scores Between Pre- and Post-Acupuncture | 1 week
  Primary outcome variables include percentage changes of EEG scores at the medial frontal gyrus, precuneus, and anterior cingulate regions from pre- to post-acupuncture at each acupuncture session. Repeated measures ANOVA used for the analysis, with fixed effects of sequence (order of acupuncture sessions), treatment (each acupuncture group), and period (1st vs 2nd session), and random patient (nested within sequence) effects included. Adjustments for multiple testing made according to the method of Westfall and Young.

SECONDARY OUTCOMES:
Symptoms of Xerostomia | 1 week
  Secondary outcomes are to determine between-acupuncture differences in radiation-induced xerostomia. Association examined between changes in neural outcomes and changes in salivary flow and self-report measures of xerostomia and other quality of life measures, controlling for the factors of acupuncture and period (1st vs 2nd) as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Cohen, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States
- Fudan University Cancer Hospital, Shanghai, China

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org